CLINICAL TRIAL: NCT03186066
Title: A Prospective Randomized Controlled Multicenter Trial for Evaluation of the Flamingo Device in Endoscopic Treatment of the Buried Bumper Syndrome.
Brief Title: Endoscopic Treatment of the Buried Bumper Syndrome: Comparison of the Flamingo Device Versus Standard Therapy
Acronym: ESCAPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kliniken Ludwigsburg-Bietigheim gGmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESCAPE
Record Dates: First submitted 2017-06-11; First posted 2017-06-14 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Buried Bumper Syndrome
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Therapy (Active Comparator): Buried Bumper Syndrome is treated by endoscopically dissecting the overgrown tissue with an endoscopic submucosal dissection knife.
  Interventions: Procedure: Standard Therapy
- Flamingo Device (Experimental): The Flamingo device is used for treatment of Buried Bumper Syndrome.
  Interventions: Device: Flamingo Device

INTERVENTIONS:
Device: Flamingo Device — Endoscopic Treatment of Buried Bumper Syndrome with the Flamingo Device
  Arms: Flamingo Device
Procedure: Standard Therapy — Endoscopic Treatment of Buried Bumper Syndrome with an endoscopic submucosal dissection knife
  Arms: Standard Therapy

SUMMARY:
Percutaneous endoscopic gastrostomy (PEG) is a method for nutrition delivery for patients with insufficient oral intake. A rare but severe complication of PEG is the Buried Bumper Syndrome (BBS). In BBS the internal fixation device of the PEG migrates along the stoma chanel. The internal fixation disc becomes covered by gastric mucosa, which causes loss of patency, fixation of the PEG and possible leakage around the PEG.

BBS can be treated endoscopically by dissecting the overgrowing tissue with endoscopic submucosal dissection (ESD) knifes. A new and alternative approach is the use of the Flamingo device, which is inserted over the PEG and then is used to radially dissect the overgrowing tissue with a cutting wire.

In this study both methods, the standard method using an ESD knife and the Flamingo device, are compared in a randomized controlled open-label trial. Primary endpoint is the time needed for PEG removal.

ELIGIBILITY:
Inclusion Criteria:

* Endoscopy proven Buried Bumper Syndrome
* PEG or Jet-PEG

Exclusion Criteria:

* Major Coagulation disorder
* Percutaneous endoscopic jejunostomy or use of a ballon fixed device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2017-06-02 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2023-04-08 (Actual)

PRIMARY OUTCOMES:
Time for Removal of PEG | Assessed at day 1 (day of intervention)

SECONDARY OUTCOMES:
Success rate | Assessed at day 1
Complications | Assessed during follow-up for up to ten days

CONTACTS AND LOCATIONS:
Locations (1):
- Klinikum Ludwigsburg, Ludwigsburg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wannhoff A, Kullmer A, Albers D, Fahndrich M, Ganten T, Wettstein M, Meier B, Schumacher B, Schmidt A, Caca K. Prospective randomized controlled trial comparing a novel and dedicated device with conventional endoscopic techniques for the treatment of buried bumper syndrome (with video). Gastrointest Endosc. 2024 Jan;99(1):23-30.e1. doi: 10.1016/j.gie.2023.07.048. Epub 2023 Aug 3. PMID 37543062